CLINICAL TRIAL: NCT06420804
Title: Evaluation of the Safety and Efficacy of an Acne Treatment Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZIIP Beauty (Industry)
Collaborators: Dermatology Consulting Services, PLLC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCS-46-20
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Mild to Moderate Acne
Keywords: Acne, Acne self care, Adult facial acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Historically Controlled Study

STUDY DESIGN:
Intervention Model Description: Single-site monadic study to evaluate the effect of a device on acne treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single-site monadic study (Experimental): Single-site monadic study to evaluate the effect of a device on acne treatment.
  Interventions: Device: ZIIP Acne Treatment Device

INTERVENTIONS:
Device: ZIIP Acne Treatment Device — Evaluation of the Safety and Efficacy of a ZIIP Acne Treatment Device
  Other Names: Historical Control

SUMMARY:
A 50-patient study in which 400 microamps of direct current was applied 3 days per week. All tolerability, safety and efficacy endpoints were met.

DETAILED DESCRIPTION:
A 50-patient study in which 400 microamps of direct current, applied 3 days per week on non-consecutive days, on all areas afflicted by acne. The results were as follow:

TOLERABILITY ASSESSMENT The tolerability endpoint was the investigator-assessed absence of skin irritation from the facial study device at any time during the 12-week study. The tolerability endpoint was met. No statistically significant skin irritation was observed by the dermatologist investigator at any time during the study.

SAFETY ASSESSMENT The safety endpoint was the absence of significant adverse reactions. No adverse reactions occurred. The safety endpoint was met.

EFFICACY ASSESSMENT The efficacy endpoint was the investigator assessed improvement in investigator global assessment (IGA) after 12 weeks of every other day device use as compared to baseline. The efficacy endpoint was met. There was a 62% reduction in inflammatory lesions and a 49% reduction in noninflammatory lesions at week 12. The IGA was reduced by 44% after 12 weeks of device use from a baseline average of 2.56 to a week 12 average of 1.42.

The ZIIP Acne Treatment Study was conducted in compliance with 21 CFR Parts 50, 56 and 812.

No protocol deviations were reported during the ZIIP Acne Treatment Study.

ELIGIBILITY:
Inclusion Criteria:

* The following represented the inclusion criteria:

  1. Subjects with mild to moderate acne (5-30 inflammatory lesions and no nodules/cysts).
  2. Male and female subjects age 18-50 years.
  3. Subjects with all Fitzpatrick skin types.
  4. Subjects of all complexion types (normal, oily, dry, combination).
  5. Subjects must have an acne lesion in all 4 zones. .
  6. Subjects who have used the same moisturizer without difficulty for 30 days and will continue using same moisturizer during the 12-week study.
  7. Subjects agree not to introduce any new colored cosmetics (lipsticks, eye shadows, facial foundations, blush, or powder).
  8. Subjects who are using no other acne products for the duration of the study.
  9. No known medical conditions that, in the investigator's opinion, may interfere with study participation.
  10. Women of childbearing potential were willing to use a form of birth control during the study. For the purpose of this study, the following are considered acceptable methods of birth control: oral contraceptives, Norplant®, Depo-Provera®, double barrier methods (e.g., condom and spermicide) and abstinence.
  11. Subjects have signed an Informed Consent Form in compliance with 21CFR, Part 50: "Protection of Human Subjects."

Exclusion Criteria:

* The following represented the exclusion criteria:

  1. Any dermatological disorder, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's skin characteristics, except for the study condition of acne.
  2. Subjects who are not willing to use the assigned study device to their face as instructed.
  3. Subjects who have used any topical prescription or OTC acne products for 2 weeks prior to study entry.
  4. Subjects who have taken any oral prescription or OTC acne products for 4 weeks prior to study entry.
  5. Subjects who have used a non-OTC cleanser without benzoyl peroxide, sulfur or salicylic acid for at least 2 weeks prior to study entry.
  6. Subject who have not had any facial treatments in the past 6 months and are willing to withhold all facial treatments during the course of the study including facials, facial peels, photo facials, laser treatments, dermabrasion, botulinum toxin (Botox), injectable filler treatments, intense pulsed light (IPL), acid treatments, tightening treatments, and/or facial plastic surgery.
  7. Subjects who are pregnant, breast feeding or planning a pregnancy.
  8. Subjects with clinically significant and/or unstable medical disorders.
  9. Subjects who are unwilling or unable to comply with the requirements of the protocol.
  10. Subjects who have a history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study.
  11. Subjects who have undergone recent facial surgery.
  12. Subjects currently participating in any other clinical trial.
  13. Subjects having started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to the study entry; or who plan on starting, stopping or changing doses of HRT or hormones for birth control during the study.
  14. Subjects who have a cardiac pacemaker, implanted defibrillator, or other implanted metallic or electronic device.
  15. Subjects who are wearing EKG monitoring equipment.
  16. Subjects with phlebitis, thrombophlebitis, broken capillaries, or varicose veins.
  17. Subjects who have seizures, epilepsy, or cancer/tumors.
  18. Subjects who have a history of hypertrophic scarring or keloid formation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-03 (Actual)

PRIMARY OUTCOMES:
Efficacy Assessment | 12 weeks
  The efficacy endpoint was the investigator assessed improvement in investigator global assessment (IGA) after 12 weeks of every other day device use as compared to baseline.

SECONDARY OUTCOMES:
Safety Assessment | 12 weeks
  The safety endpoint was the absence of significant adverse reactions. No adverse reactions occurred.

OTHER OUTCOMES:
Tolerability Assessment | 12 weeks
  The tolerability endpoint was the investigator-assessed absence of skin irritation from the facial study device at any time during the 12-week study.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe D Draelos, MD, Principal Investigator — Lead Investigator
Locations (1):
- ZIIP Beauty, Pleasant Hill, California, United States

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan to share IPD data

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT06420804/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT06420804/ICF_001.pdf